CLINICAL TRIAL: NCT04036812
Title: Ultrasound Guided Superficial Cervical Plexus Block for Analgesia After Craniotomy Via Suboccipital Retrosigmoid Approach: A Randomized Controlled Trial
Brief Title: Superficial Cervical Plexus Block for Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Associate professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-06-29
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Plexus Block;Analgesia;Neurosurgery
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superficial cervical plexus block group (Experimental)
  Interventions: Procedure: Superficial cervical plexus block
- Control group (Sham Comparator)
  Interventions: Other: Control group

INTERVENTIONS:
Procedure: Superficial cervical plexus block — superficial cervical plexus nerve block will be performed under the guidance of ultrasound
  Arms: Superficial cervical plexus block group
Other: Control group — ultrasound guidance will be used to determine the location of superficial cervical plexus nerve. The puncture will also be performed by ultrasound guidance, covered with opaque infusion dressing but performed with infusion of 10 ml normal saline.
  Arms: Control group

SUMMARY:
The incidence of postoperative pain after craniotomy is high. Severe postoperative pain can lead to a series of complications that are detrimental to the recovery of craniotomy patients. Compound local scalp nerve block is a good choice for analgesia after craniotomy. However, the scalp nerve block commonly cannot cover the area of suboccipital retrosigmoid approach craniotomy, leading to incomplete block. Superficial cervical plexus block (SCPB) is theoretically promising to solve the analgesia requirements of such surgical approach. At the same time, ultrasound guidance can not only accurately locate, ensure the effect of block and avoid accidental injury during puncture. The purpose of this study is to explore whether ultrasound-guided superficial cervical plexus block can safely and effectively reduce the requirement of analgesic drugs and pain after craniotomy via suboccipital retrosigmoid approach.

ELIGIBILITY:
Inclusion Criteria:

1. Elective suboccipital retrosigmoid approach approach craniotomy;
2. Age between 18 and 65 years;
3. American Society of Anesthesiologists (ASA) physical status I-III.

Exclusion Criteria:

1. The patients or legal clients refuse to provide informed consent;
2. Local infection;
3. Preoperative impairment of consciousness and cognitive function;
4. Uncontrolled hypertension;
5. Inability to communicate;
6. Allergies to experimental drugs;
7. History of drug abuse;
8. History of chronic headache;
9. Aphasia and hearing impairment;
10. Patients undergoing second craniotomy;
11. Body mass index < 18.5 kg/m2 or > 35.0 kg/m2;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
the cumulative consumption of sufentanil by the PCA | 24 hours after surgery
  the cumulative consumption of sufentanil by the PCA 24 hours after surgery

SECONDARY OUTCOMES:
Use of analgesics by the PCA after operation | at 1, 2, 4, 48 hours after surgery.
  the cumulative consumption of sufentanil by PCA
Pain severity score | at 1, 2, 4, 24, 48 hours after surgery
  It will be accessed using NRS
Anesthesia recovery quality score： | at 1 hour after surgery
  It will be accessed at postoperative 1 and 2 hours using the Anesthesia Steward Emergence Scale. The Anesthesia Steward Emergence Scale(0-6) is divided into three parts: the degree of wakefulness - 2 points for complete recovery, 1 point for response to stimulation, 0 point for no response to stimulation; the degree of airway patency - 2 points for cough according to the doctor's order, 1 point for maintenance of airway patency without support, 0 point for support required for respiratory tract; 2 points for conscious activities of limbs with limb mobility, 1 point for unconscious activities of limbs, point for no activities of limbs.
Patient analgesic satisfaction | at 24 hours after surgery
  Patient satisfaction with overall pain management will be evaluated at 24 hours after surgery using NRS

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Peng, M.D., Principal Investigator — Beijing Tian Tan Hospital, Capital Medical University
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Beijing TianTan Hospital, Beijing

REFERENCES:
- [Derived] Zeng M, Li R, Xu X, Wang D, Dong J, Li S, Kass IS, Peng Y, Jia W. Ultrasound-guided superficial cervical plexus block reduces opioid consumption in patients undergoing craniotomy via suboccipital retrosigmoid approach: a randomized controlled trial. Reg Anesth Pain Med. 2022 Jun 29:rapm-2022-103534. doi: 10.1136/rapm-2022-103534. Online ahead of print. PMID 35768167
- [Derived] Peng K, Zeng M, Dong J, Yan X, Wang D, Li S, Peng Y. Ultrasound-guided superficial cervical plexus block for analgesia in patients undergoing craniotomy via suboccipital retrosigmoid approach: study protocol of a randomised controlled trial. BMJ Open. 2020 Feb 5;10(2):e034003. doi: 10.1136/bmjopen-2019-034003. PMID 32029493